CLINICAL TRIAL: NCT01238016
Title: Evaluation of Hypo-Safe Hypoglycaemia Alarm Device - a Pilot Study - A One Month Non-controlled Observational Study
Brief Title: Evaluation of Hypo-Safe Hypoglycaemia Alarm Device - a Pilot Study
Acronym: Pilot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Replaced by new study
Sponsor: UNEEG Medical A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H01A03
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- device (Other): Device implant and EEG recording
  Interventions: Device: experimental

INTERVENTIONS:
Device: experimental

SUMMARY:
The trial aims at measuring the safety and performance of the Hyposafe device.

DETAILED DESCRIPTION:
Safety: To evaluate safety issues related to implantation and use of the Hyposafe hypoglycaemia alarm device Performance: To evaluate the stability of the hypoglycaemia alarm device.

ELIGIBILITY:
Inclusion Criteria:

Healthy control subjects or and

* Male and female patient with type 1 diabetes for at least one year
* Age 18-70 years
* Impaired awareness of hypoglycaemia as defined by

  * A score of ≥4 on the Gold-scale or
  * Two or more occasions of severe hypoglycaemia (need of help from third person) within the past 12 month
* Multiple injection insulin therapy or continuous insulin injection therapy
* For female participants: Not pregnant and, if child bearing potential, usage of reliable anti-contraceptive method during the study period

Exclusion Criteria:

* Severe cardiac disease

  * History of myocardial infarction
  * Cardiac arrhythmia
* Previous stroke or cerebral haemorrhage and any other structural cerebral disease
* Active cancer or cancer diagnosis within the past five years
* Uremia defined as s-creatinine above 3 times upper reference value
* Liver disease defined as s-ALAT above 3 times upper reference interval
* Inability to understand the informed consent
* Epilepsy
* Use of antiepileptic drugs for any purposes
* Clinical important hearing impairment
* Use of active implantable medical device including

  * Pacemaker and ICD-unit
  * Cochlear implant
* Use of following drugs

  * Chemotherapeutic drugs of any kind
  * Methotrexate
  * Third generation antipsychotic drugs (aripiprazole, quetiapine, clozapine, ziprasidone, paliperidone, risperidone, sertindole, amisulpride, olanzapine)
* Abuse of alcohol (defined as consumption of > 250g alcohol (in Danish: 21 "genstande") per week or abuse of any other neuroactive substances
* Infection at the site of device-implantation
* Any hemorrhagic disease
* Diving (snorkel diving allowed) or parachute jumping
* Patients that are judged incapable of understanding the patient information or who are not capable of carrying through the investigation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Device performance | End of observation

CONTACTS AND LOCATIONS:
Locations (1):
- Esbjerg Sygehus, Esbjerg, Denmark